CLINICAL TRIAL: NCT04417946
Title: Peer-led Social Media Intervention to Prevent HIV Among Young Men Who Have Sex With Men (YMSM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000022728; 1H79TI080736 (Other Grant/Funding Number: Substance Abuse and Mental Health Services Administration)
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pre-Exposure Prophylaxis; Hiv; Men
Keywords: pre-exposure prophylaxis (PrEP); social media intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Messages (Experimental): The peer leaders and the study staff will post PrEP related health messages
  Interventions: Behavioral: PrEP messages
- Health messages (Active Comparator): The peer leaders and study staff will post general health messages that are not related to sexual health.
  Interventions: Behavioral: Heath messages

INTERVENTIONS:
Behavioral: PrEP messages — The peer leaders and the study staff will post PrEP related health messages
  Arms: PrEP Messages
Behavioral: Heath messages — The peer leaders and study staff will post general health messages that are not related to sexual health
  Arms: Health messages

SUMMARY:
The aim of this study is to examine the effect of social media intervention on the use of pre-exposure prophylaxis (PrEP) by young men who have sex with men (YMSM) in the greater New Haven area.

DETAILED DESCRIPTION:
There are three specific aims of this study. In the first specific aim, two focus group discussions (FGDs) of YMSM will be conducted to assess the feasibility and acceptability of social media intervention. In the second specific aim of the study, a quasi-pre-post experimental study will be conducted to examine the effect of social media intervention on PrEP uptake (primary outcome) and PrEP use intention, HIV testing, PrEP knowledge, self-efficacy and social support (secondary outcome). In the third specific aim of the study, the most important topics around PrEP will be assessed on the Facebook page of the intervention group by conducting a content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male or transgender man
* Self-identification as gay or bi-sexual
* Resident of greater New Haven area
* Willing and able to use Facebook during the span of the study

Exclusion Criteria:

* • Women will not be included in the study

  * Under the age of 18 and over the age of 29
  * Unable to provide informed consent
  * Verbally or physically threatening to research staff

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biologically male or transgender man
Enrollment: 227 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
PrEP uptake | PrEP uptake at baseline
  Actual PrEP uptake: participants self report if they use prep (Yes/No)
PrEP uptake | PrEP uptake (Yes/No) at 24-weeks
  Actual PrEP uptake: participants self report if they use prep (Yes/No)

SECONDARY OUTCOMES:
HIV testing | baseline
  Date of the last HIV test: participants self report the date of their last HIV test as a function of time in days.
HIV testing | 24-weeks
  Date of the last HIV test: participants self report the date of their last HIV test as a function of time in days.
PrEP use intention | PrEP use intention at baseline
  Willingness to use/likelihood of using PrEP in the next 6 months : self reported assessment to measure participants' willingness to use prep in the next 6 month s on a single question using Likert scale from 1(very unlikely) to 7 (very likely)
PrEP use intention | PrEP use intention at 24-weeks
  Willingness to use/likelihood of using PrEP in the next 6 months : self reported assessment to measure participants' willingness to use prep in the next 6 month s on a single question using Likert scale from 1(very unlikely) to 7 (very likely)
PrEP knowledge | PrEP knowledge at baseline
  Knowledge of PrEP for HIV prevention: self reported assessment to measure participants' knowledge on PrEP on a set of True or False questions
PrEP knowledge | PrEP knowledge at 24-weeks
  Knowledge of PrEP for HIV prevention: self reported assessment to measure participants' knowledge on PrEP on a set of True or False questions
self efficacy to use PrEP | self efficacy to use PrEP at baseline
  Beliefs in his/her ability of using PrEP: participants self report their level of confidence in taking PrEP on a set of items using Likert scales from 1 (Not at all confident) to 5 (completely confident)
self efficacy to use PrEP | self efficacy to use PrEP at 24-weeks
  Beliefs in his/her ability of using PrEP: participants self report their level of confidence in taking PrEP on a set of items using Likert scales from 1 (Not at all confident) to 5 (completely confident)
motivation to use PrEP | motivation to use PrEP at baseline
  How motivated s/he is to use PrEP and what motivates s/he to use PrEP: self reported assessment to measure participants' different types of motivation to use PrEP on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)
motivation to use PrEP | motivation to use PrEP at 24-weeks
  How motivated s/he is to use PrEP and what motivates s/he to use PrEP: self reported assessment to measure participants' different types of motivation to use PrEP on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)
PrEP stigma | PrEP stigma at baseline
  Perceived stigma related to PrEP use: self reported assessment to measure perception of stigma related to PrEP use on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)
PrEP stigma | PrEP stigma at 24-weeks
  Perceived stigma related to PrEP use: self reported assessment to measure perception of stigma related to PrEP use on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)
Social support for PrEP use | Social support for PrEP use at baseline
  Help and support that individuals receive that can facilitate PrEP uptake: Perceived stigma related to PrEP use: self reported assessment to measure perception of social support related to PrEP use on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)
Social support for PrEP use | Social support for PrEP use at 24-weeks
  Help and support that individuals receive that can facilitate PrEP uptake: Perceived stigma related to PrEP use: self reported assessment to measure perception of social support related to PrEP use on a set of items using Likert scales from 1(strongly disagree) to 7 (strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, M.D., M.A., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - APNH: A Place to Nourish your Health (APNH), New Haven, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
All data will be kept confidential.